CLINICAL TRIAL: NCT02548208
Title: Effect of a Single Administration of Focused Extracorporeal Shock Wave in the Relief of Delayed-Onset Muscle Soreness
Brief Title: Single Focused Shock Wave in the Release od Delayed Onset Muscle Soreness (DOMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Johannes Fleckenstein (Other)
Responsible Party: Sponsor-Investigator, Dr. Johannes Fleckenstein, Senior Researcher, Goethe University
Organization: Goethe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESWT_DOMS
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Musculoskeletal Pain; Athletic Injuries
MeSH Terms: conditions — Musculoskeletal Pain; Athletic Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Verum focused extracorporeal shockwave therapy (Active Comparator): Verum focused extracorporeal shockwave therapy is applied at 7 equidistant points, perpendicular to the belly of the biceps brachii muscle on a thought line between the radial tuberosity and the coracoid process (Dermagold120, Tissue Regeneration Technologies, Woodstock, Georgia, U.S.). Shock waves are generated by electrohydraulic mechanisms.
  Interventions: Device: Verum focused extracorporeal shockwave
- Sham shock wave (Sham Comparator): Sham shock wave is performed using the same device as stated above, but using a special applicator that has been isolated with layers of metal and water by the manufacturer, extinguishing the transmitted energy. The study personal is blinded to the applicators. All handling, adjustments and noises are thus same in this group.
  Interventions: Device: Sham shock wave
- Control (No Intervention): Control procedure stipulates participants to lay down on the same therapy table for 5 minutes receiving no intervention.

INTERVENTIONS:
Device: Verum focused extracorporeal shockwave — the concentrated shockwave energy per unit area (energy flux density EFD) can vary from 0.06 to 0.09 mJ/mm2. The pulse ratio per point is 200.
  Other Names: focused extracorporeal shockwave therapy
  Arms: Verum focused extracorporeal shockwave therapy
Device: Sham shock wave — Sham shock wave is performed using the same device as stated above, but using a special applicator that has been isolated with layers of metal and water by the manufacturer, extinguishing the transmitted energy.
  Arms: Sham shock wave

SUMMARY:
The study is a single-center, double blinded, randomized controlled trial aimed to investigate the effects of focused extracorporeal shockwave therapy (fESWT) on Delayed Onset Muscle Soreness (DOMS) of the non-dominant biceps brachialis muscle in healthy voluntary adults.

DETAILED DESCRIPTION:
Forty-five participants agreed to participate and signed a written informed consent. After enrollment, muscle soreness was induced and participants were subsequently randomized to receive either (1) focused extracorporeal shockwave therapy (Verum), (2) sham shock wave (Sham) or (3) no treatment (Control). Thereafter, treatments were administered once, only. Measures were repeated after the treatment and at 24, 48 and 72 hours. Main outcome parameter was the pain intensity at rest and in movement as assessed by visual analogue scale (VAS) in the elbow region of the non-dominant arm. Secondary outcome included the pressure pain threshold (PPT) over the biceps muscle belly, the maximum isometric voluntary force (MIVF) of the elbow flexors and the assessing the impairment of activities of the daily living. Participants were followed-up 72 hours after the induction of Delayed Onset Muscle Soreness.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 18+
* voluntariness

Exclusion Criteria:

* pain
* pregnancy
* musculoskeletal disease
* systemic neurological disease
* cancer
* coagulation disorder
* mental illness
* drug addiction
* allergy to the ultrasound gel
* cardiac illness
* vascular disease of the limbs or the central nervous system
* regional scars
* regional skin transplants or hypoesthesia
* allergic or other forms of acute dermatitis
* chronic intake of analgesic, neuroleptics, antidepressants, corticoids or alpha2-blockers
* current state of delayed onset muscle soreness
* extracorporeal shockwave therapy within last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 72 hours
  Pain intensity at the elbow region during active movement of the biceps muscle is assessed using a visual analogue scale (VAS) ranging from 0 to 10 cm (with 0 indicating no pain and 10 experiencing the worst imaginable pain).

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | 72 hours
  PPT is assessed using a mechanical pressure algometer (pdt, Rome, Italy) with increasing force at a rate of approximately 1 kg/cm2/s until the participant reported a painful sensation; and the force value is recorded (kg/cm2).
Maximum isometric voluntary force MIVF | 72 hours
  MIVF is easured using a strain-gauge force transducer (ASYS® SPOREG, Offenbach, Germany). Peak strength values (N) are recorded.
Activities of daily living (ADL) | 72 hours
  This test comprises the asssessment of the impairment of six complex movements (each on a VAS 0-10 cm) and the mean VAS of all items is kept to describe the impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Banzer, Prof, Study Director — Department of Sports Medicine, Institute of Sports Sciences, Goethe-University Frankfurt, Germany
Locations (1):
- Department of Sports Medicine, Institute of Sports Sciences, Goethe University, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Fleckenstein J, Friton M, Himmelreich H, Banzer W. Effect of a Single Administration of Focused Extracorporeal Shock Wave in the Relief of Delayed-Onset Muscle Soreness: Results of a Partially Blinded Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 May;98(5):923-930. doi: 10.1016/j.apmr.2016.11.013. Epub 2016 Dec 16. PMID 27993588